CLINICAL TRIAL: NCT04957212
Title: A Phase III, Randomized, Two-armed, Parallel, Triple-blind, Active-controlled, Equivalency Clinical Trial of Efficacy and Safety Pertuzumab® (CinnaGen Co.) Compared With Perjeta® (Originator Pertuzumab) in Neoadjuvant Treatment of HER2+ Breast Cancer
Brief Title: Comparing Efficacy and Safety Between Pertuzumab® and Perjeta® in Neoadjuvant Treatment of HER2+ Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PER.CIN.BN.95.III
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: HER2-positive Breast Cancer
Keywords: Pertuzumab; HER2-positive Breast Cancer; Neoadjuvant treatment; Equivalency clinical trial
MeSH Terms: interventions — Trastuzumab; pertuzumab; Carboplatin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly assigned to treatment by a central randomization procedure via telephone call for each consecutive eligible patient. Randomization codes were allocated after all eligibility criteria were approved, stratification factors were identified and the informed consent form was signed.
  After randomization procedure, a code was allocated to each patient that was used as patient identifier throughout the study. The assigned code was denoted by 4 initials (corresponding to the 2 first letter of the first name, the 2 first letter of the first surname) and 3 numbers (center code).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCHP regimen (trastuzumab, pertuzumab® (CinnaGen Co.), carboplatin, and docetaxel) (Experimental): Study drugs are administered intravenously on a 3-weekly schedule and given consecutively on the same day in the following sequence: trastuzumab, followed by pertuzumab, carboplatin, and docetaxel. Trastuzumab is given at an initial dose of 8 mg/kg, followed by 6 mg/kg; pertuzumab® (CinnaGen Co.) is given at an initial dose of 840 mg, followed by 420 mg. Carboplatin is administered at a dose of AUC6 (area under the plasma concentration-time curve) and docetaxel is given at 75 mg/m2.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin; Drug: Docetaxel
- TCHP regimen (trastuzumab, Perjeta®, carboplatin, and docetaxel) (Active Comparator): Study drugs are administered intravenously on a 3-weekly schedule and given consecutively on the same day in the following sequence: trastuzumab, followed by pertuzumab, carboplatin, and docetaxel. Trastuzumab is given at an initial dose of 8 mg/kg, followed by 6 mg/kg; Perjeta® is given at an initial dose of 840 mg, followed by 420 mg. Carboplatin is administered at a dose of AUC6 (area under the plasma concentration-time curve) and docetaxel is given at 75 mg/m2.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab — An initial dose of 8 mg/kg, followed by 6 mg/kg every 3-weeks
Drug: Pertuzumab — An initial dose of 840 mg, followed by 420 mg every 3-weeks
Drug: Carboplatin — A dose of AUC6 (area under the plasma concentration-time curve) every 3-weeks
Drug: Docetaxel — 75 mg/m2 every 3-weeks

SUMMARY:
This study was a phase III, multicenter, triple-blind, equivalency clinical trial to determine the therapeutic efficacy and safety between Pertuzumab® (CinnaGen Co.) compared to originator pertuzumab in HER2-positive early breast cancer patients.

Patients were stratified dynamically for random assignment to treatment with either Pertuzumab® (CinnaGen Co.) or originator pertuzumab, and received neoadjuvant TCHP regimen every 3- weeks.

DETAILED DESCRIPTION:
This study was a phase III, multicenter, triple-blind , equivalency clinical trial to determine the therapeutic efficacy and safety between Pertuzumab® (CinnaGen Co.) compared to originator pertuzumab in HER2-positive early breast cancer patients.

Patients stratified dynamically according to two factors: type of breast cancer (inflammatory, locally and operable) and estrogen/ progesterone receptor (ER/PR) (positive or negative) with 1:1 allocation ratio.

Study drugs were administered intravenously on a 3-weekly schedule and were given consecutively on the same day in the following sequence: trastuzumab, followed by pertuzumab, carboplatin, and docetaxel (TCHP regimen).

The primary endpoint was breast pCR (bpCR). Secondary efficacy endpoints included total pCR (tpCR); objective response rate (ORR) and rate of breast-conserving surgery (BCS) for patients for whom mastectomy was planned before treatment (T2-3).

During this study, adverse events (AEs) were monitored continuously. As an adverse event of special interest (AESI), left ventricular ejection fraction (LVEF) decreased was monitored and assessed by echocardiography throughout the study. Immunogenicity was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70 years.
* Diagnosed with locally advanced (T2-3, N2-3, M0 or T4a-c, any N, M0), inflammatory (T4d, any N, M0) or operable (T2-3, N0-1, M0), invasive breast cancer.
* Primary tumor > 2 cm in diameter.
* HER2 positive breast cancer confirmed (Tumors must be IHC 3+ or FISH/CISH + for IHC 2+ tumors).
* Baseline LVEF ≥ 55% measured by echocardiography.
* Performance status ECOG ≤ 1
* Signed informed consent.

Exclusion Criteria:

* Metastatic disease (Stage IV) or bilateral breast cancer.
* Previous anticancer therapy or radiotherapy for any malignancy.
* Other malignancy, except for carcinoma in situ of the cervix or basal cell carcinoma.
* Received any investigational treatment within 4 weeks of study start.
* At least 4 weeks since major surgery.
* Uncontrolled hypertension (systolic > 150 and/or diastolic > 100), unstable angina, CHF of any NYHA classification, serious cardiac arrhythmia requiring treatment, history of myocardial infarction within 6 months of enrollment.
* Hematological, biochemical and organ dysfunction:

  1. Inadequate bone marrow function: Absolute Neutrophil Count (ANC) < 1500 cells/ µL, Platelet count < 100,000 cells/ µL and Hb < 9 g/dL).
  2. Impaired liver function: serum [total] bilirubin > 1.25 x ULN, AST/ALT > 1. 5 x ULN with ALP > 2.5 x ULN
  3. Inadequate renal function: serum creatinine > 1.5 x ULN.
* Dyspnea at rest or other diseases which require continuous oxygen therapy.
* Severe uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, metabolic, etc).
* Current chronic daily treatment with corticosteroids (dose of ≥10 mg Oral prednisolone, or equivalent [excluding inhaled steroids])
* Subjects with known infection with HIV, HBV, and HCV.
* Known hypersensitivity to any of the study drugs or excipients.
* Pregnant and/or lactating women or subjects with reproductive potential not willing to use effective methods of contraception.
* Subjects assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol (e.g.: physical, psychological and mental problems)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 214 (Actual)
Dates: Start 2018-08-11 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Behrouz Najafi, MD, Principal Investigator — Assistant Professor of Hematology and Oncology Research Center
Locations (44):
- Iran (44):
  - Besat Clinic, Rasht, Gilan Province
  - Dr. Behrouz Najafi's office, Rasht, Gilan Province
  - Dr. Mehdi Mirblouk's office, Rasht, Gilan Province
  - Razi Hospital, Rasht, Gilan Province
  - Dr. Aboulqasem Allahyari's office, Mashhad, Khorasan Razavi
  - Imam Reza Hospital, Mashhad, Khorasan Razavi
  - Qaem Hospital, Mashhad, Khorasan Razavi
  - Sanabad Hospital, Mashhad, Khorasan Razavi
  - Arvand Hospital, Ahvāz, Khozestan
  - Baqaei Hospital, Ahvāz, Khozestan
  - Shafa Hospital, Ahvāz, Khozestan
  - Milad Hospital, Isfahan
  - Saba Clinic, Isfahan
  - Seyed-Al-Shohada Hospital, Isfahan
  - Sheikh Mofid Clinic, Isfahan
  - Dr. Behjat Kalantari's office, Kerman
  - Javad-Al-Aemeh Clinic, Kerman
  - Shahid Bahonar Hospital, Kerman
  - Dr. Mehrdad Payende's office, Kermanshah
  - Amir Hospital, Shiraz
  - Namazi Hospital, Shiraz
  - Shahid Faghihi Hospital, Shiraz
  - Shams Hospital, Tabriz
  - Baqiatallah Hospital, Tehran
  - BuoAli Hospital, Tehran
  - Dr. Safa Najjar Najafi's office, Tehran
  - Ebn-Sina Hospital, Tehran
  - Firoozgar Hospital, Tehran
  - Imam Khomeini Hospital, Tehran
  - Iran-Mehr Hospital, Tehran
  - Jam Hospital, Tehran
  - Jihad University Clinic, Tehran
  - Masih Daneshvari Hospital, Tehran
  - Massoud Clinic, Tehran
  - Mehrad Hospital, Tehran
  - Naft Hospital, Tehran
  - Rasool Akram Hospital, Tehran
  - Resalat Hospital, Tehran
  - Sajjad Hospital, Tehran
  - Sina Hospital, Tehran
  - Taleghani Hospital, Tehran
  - Tehran Hospital, Tehran
  - Toos Hospital, Tehran
  - Dr.Mortazavizadeh's office, Yazd

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Started | 107 | 107
Completed | 107 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel) | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.56 (10.31) | 44.35 (9.81) | 45.95 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 107 | 107 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.27 (5.30) | 27.27 (4.38) | 27.77 (4.87)
BSA [Mean (Standard Deviation); unit: m^2] | 1.79 (0.18) | 1.79 (0.18) | 1.79 (0.18)
IHC2+ [Count of Participants; unit: Participants]
  FISH+ | 3 | 3 | 6
  CISH+ | 6 | 3 | 9
IHC3+ [Count of Participants; unit: Participants] | 98 | 101 | 199
ER/PR+ [Count of Participants; unit: Participants] | 63 | 64 | 127
ER/PR- [Count of Participants; unit: Participants] | 44 | 43 | 87
Type of breast cancer [Count of Participants; unit: Participants]
  Inflammatory | 6 | 6 | 12
  Locally advanced | 49 | 48 | 97
  Operable | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Breast Pathological Complete Response (bpCR)
Description: bpCR defined as the absence of invasive neoplastic cells in the breast at microscopic examination of the primary tumor at surgery following primary systemic therapy (ypT0/is)
Time Frame: 18-20 weeks after first intervention
Measure: Count of Participants; unit: Participants
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Number analyzed (Participants) | 105 | 102
Participants | 71 | 73
Statistical Analysis 1: Comparison: TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) vs TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel); Test type: Equivalence — We used an equivalence margin of 0.2 for the primary endpoint; p = 0.54, Chi-squared; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.16 to 0.09]

2. Secondary Outcome: Total Pathological Complete Response (tpCR)
Description: tpCR defined as no invasive tumor residues in the breast and lymph nodes (ypT0/is ypN0)
Time Frame: 18-20 weeks after first intervention
Measure: Count of Participants; unit: Participants
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Number analyzed (Participants) | 107 | 107
Participants | 60 | 68
Statistical Analysis 1: Comparison: TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) vs TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel); Test type: Other; p = 0.26, Chi-squared; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.21 to 0.06]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR defined as the proportion of patients who achieved a complete or partial response
Time Frame: 18-20 weeks after first intervention
Measure: Count of Participants; unit: Participants
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Number analyzed (Participants) | 107 | 107
Participants
  Complete Response | 64 | 61
  Partial Response | 30 | 29
  Progressive Disease | 2 | 3
  Stable Disease | 3 | 2
  Unknown | 8 | 12
Statistical Analysis 1: Comparison: TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) vs TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel); Test type: Other; p = 0.99, Fisher Exact

4. Secondary Outcome: Rate of Breast-conserving Surgery (BCS)
Description: Rate of BCS for patients for whom mastectomy was planned before treatment (T2-3)
Time Frame: 18-20 weeks after first intervention
Measure: Count of Participants; unit: Participants
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Number analyzed (Participants) | 64 | 59
Participants
  Lumpectomy | 20 | 21
  Mastectomy | 44 | 37
  Unknown | 0 | 1
Statistical Analysis 1: Comparison: TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) vs TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel); Test type: Other; p = 0.56, Chi-squared

5. Secondary Outcome: Safety Assessment Including Treatment Related Adverse Events
Description: Safety assessment, including the incidence of all reported AEs and abnormal laboratory results was done. All AEs were classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events were graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs was assessed according to International Council for Harmonization (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.
Time Frame: Throughout the study duration (from first visit to week 18-20)
Population: A total of 214 patients were analyzed for AEs.Reports were based on the Safety set. The safety set included all randomized patients who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel): Study drugs are administered intravenously on a 3-weekly schedule and given consecutively on the same day in the following sequence: trastuzumab, followed by pertuzumab, carboplatin, and docetaxel. Trastuzumab is given at an initial dose of 8 mg/kg, followed by 6 mg/kg; pertuzumab® (CinnaGen Co.) is given at an initial dose of 840 mg, followed by 420 mg. Carboplatin is administered at a dose of AUC6 (area under the plasma concentration-time curve) and docetaxel is given at 75 mg/m2.
  Trastuzumab: An initial dose of 8 mg/kg, followed by 6 mg/kg every 3-weeks Pertuzumab: An initial dose of 840 mg, followed by 420 mg every 3-weeks Carboplatin: A dose of AUC6 (area under the plasma concentration-time curve) every 3-weeks Docetaxel: 75 mg/m2 every 3-weeks
- TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetax: Study drugs are administered intravenously on a 3-weekly schedule and given consecutively on the same day in the following sequence: trastuzumab, followed by pertuzumab, carboplatin, and docetaxel. Trastuzumab is given at an initial dose of 8 mg/kg, followed by 6 mg/kg; Perjeta® is given at an initial dose of 840 mg, followed by 420 mg. Carboplatin is administered at a dose of AUC6 (area under the plasma concentration-time curve) and docetaxel is given at 75 mg/m2.
  Trastuzumab: An initial dose of 8 mg/kg, followed by 6 mg/kg every 3-weeks Pertuzumab: An initial dose of 840 mg, followed by 420 mg every 3-weeks Carboplatin: A dose of AUC6 (area under the plasma concentration-time curve) every 3-weeks Docetaxel: 75 mg/m2 every 3-week
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetax
Number analyzed (Participants) | 107 | 107
Participants | 107 | 107

6. Secondary Outcome: Abnormal Laboratory Data
Description: Laboratory data including CBC diff have been assessed. All abnormal values were recorded as adverse event.
Time Frame: Throughout the study duration (from first visit to week 18-20)
Reporting Status: Not Posted

7. Secondary Outcome: Decrease in Left Ventricular Ejection Fraction (LVEF)
Description: LVEF decrease was measured by echocardiography. All cases with a decrease more than 10% from baseline which meet <50%, will be recorded as adverse events.
Time Frame: every 6 week (from first visit to week 18-20)
Reporting Status: Not Posted

8. Secondary Outcome: Incidence of Symptomatic Left Ventricular Systolic Dysfunction (LVSD)
Description: In this study, LVSD was evaluated by measuring the decrease in LVEF (outcome measure 5) and assessing the clinical symptoms of the study participants based on physician opinion.
Time Frame: Throughout the study duration (from first visit to week 18-20)
Reporting Status: Not Posted

9. Secondary Outcome: Immunogenicity
Description: The enzyme-linked immunosorbent assay (ELISA) method was used for the assessment of anti-drug antibodies (ADAs).
Time Frame: Every 3 weeks (from first intervention to week 18)
Population: A total of 214 patients were analyzed for immunogenicity assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
Number analyzed (Participants) | 107 | 107
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 18-20 weeks
Arm/Group | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 24/107 | 15/107
Other Adverse Events (participants affected / at risk) | 107/107 | 104/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) (N=107) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel) (N=107)
Dyspnoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 14 (19) | 10 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Fatty liver (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCHP Regimen (Trastuzumab, Pertuzumab® (CinnaGen Co.), Carboplatin, and Docetaxel) (N=107) | TCHP Regimen (Trastuzumab, Perjeta®, Carboplatin, and Docetaxel) (N=107)
Anaemia (Blood and lymphatic system disorders) | 103 (443) | 100 (477)
Thrombocytopenia (Blood and lymphatic system disorders) | 68 (185) | 69 (201)
Nausea (Gastrointestinal disorders) | 64 (114) | 71 (139)
Diarrhoea (Gastrointestinal disorders) | 60 (107) | 67 (122)
Leukopenia (Blood and lymphatic system disorders) | 56 (127) | 51 (100)
Neutropenia (Blood and lymphatic system disorders) | 49 (95) | 47 (101)
Vomiting (Gastrointestinal disorders) | 46 (82) | 53 (82)
Abdominal pain (Gastrointestinal disorders) | 43 (66) | 37 (51)
Pain (General disorders) | 38 (49) | 33 (42)
Dyspepsia (Gastrointestinal disorders) | 37 (51) | 31 (52)
Aphthous ulcer (Gastrointestinal disorders) | 12 (12) | 7 (7)
Constipation (Gastrointestinal disorders) | 16 (30) | 20 (24)
Dysgeusia (Gastrointestinal disorders) | 9 (11) | 8 (9)
Stomatitis (Gastrointestinal disorders) | 18 (18) | 10 (11)
Asthenia (General disorders) | 35 (45) | 26 (42)
Chest pain (General disorders) | 7 (7) | 7 (8)
Chills (General disorders) | 13 (13) | 7 (8)
Decreased appetite (General disorders) | 30 (40) | 31 (38)
Fatigue (General disorders) | 22 (28) | 13 (16)
Flushing (General disorders) | 11 (14) | 6 (7)
Mucosal inflammation (General disorders) | 8 (8) | 9 (10)
Oedema (General disorders) | 8 (8) | 4 (4)
Oedema peripheral (General disorders) | 9 (12) | 10 (14)
Pyrexia (General disorders) | 7 (8) | 14 (17)
Nasopharyngitis (Infections and infestations) | 11 (12) | 14 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 18 (22) | 17 (27)
Dizziness (Nervous system disorders) | 18 (25) | 11 (11)
Headache (Nervous system disorders) | 11 (13) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 9 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (23) | 16 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (23) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 21 (25) | 26 (35)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 6 (9) | 5 (9)
Xeroderma (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Epistaxis (Vascular disorders) | 13 (14) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04957212/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04957212/SAP_001.pdf